CLINICAL TRIAL: NCT00173407
Title: Correlation of PTEN and IGFBP-3 in the Invasion of Ovarian Endometrioid Carcinoma
Brief Title: PTEN and IGFBP-3 Correlation in Ovarian Carcinoma Invasion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9461700640
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian endometrioid carcinoma; invasion; IGFBP-3; transfection; signal transduction; PTEN; methylation
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Methylation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: immunohistochemical, methylation, gene transfection

SUMMARY:
We have identified insulin-like growth factor binding protein (IGFBP)-3 as an invasion suppressor gene in ovarian endometrioid carcinoma, and showed association with lower cancer migration, invasion and metastasis. Recently, a novel model of ovarian EC formation from endometriosis was reported, and PTEN was found to be a major protein involved. Inactivation of PTEN has been reported in some ovarian EC tumors and methylation was suggested as one of the major epigenetic changes. This tumorigenesis model has lots of similarity to our established invasion model. Therefore, we plan to study the important of PTEN expression in ovarian EC and if inactivation of PTEN and IFGBP-3 is through methylation. Furthermore, by studying the signal transduction pathways using PTEN and IGFBP-3 transfection, we plan to study the mutual interaction between PTEN and IGFBP-3 on the suppression of tumor invasion in ovarian EC.

DETAILED DESCRIPTION:
We have successfully established an ovarian cancer cell line (OVTW-59), which was derived from an ovarian endometrioid carcinoma (EC), and have also established an ovarian EC invasion model. By using cDNA microarray and quantitative reverse-transcriptase polymerase chain reaction, we identified insulin-like growth factor binding protein (IGFBP)-3 as an invasion suppressor gene, which were associated with lower cancer migration, invasion and metastasis. Clinically, lower IGFBP-3 was found associated with significantly higher tumor grade, advanced stage and poor survival in patients with EC tumors. Furthermore, we have proved IGFBP-3 expression correlated with lower Erk activation, but with no effect on the activation of Akt. All these two signal transduction proteins have crucial roles in cancer invasion. Recently, a novel model of ovarian EC formation from endometriosis was reported, and PTEN was found to be a major protein involved. Inactivation of PTEN has been reported in some ovarian EC tumors and methylation was suggested as one of the major epigenetic changes. This tumorigenesis model has lots of similarity to our established invasion model. Therefore, we plan to study the important of PTEN expression in ovarian EC and if inactivation of PTEN and IFGBP-3 is through methylation. Furthermore, by studying the signal transduction pathways using PTEN and IGFBP-3 transfection, we plan to study the mutual interaction between PTEN and IGFBP-3 on the suppression of tumor invasion in ovarian EC.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of ovarian endometrioid carcinoma

Exclusion Criteria:

other types of ovarian epithelial carcinoma

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
migration
invasion
metastasis

SECONDARY OUTCOMES:
Immunohistochemical staining
methylation
signal tranduction

CONTACTS AND LOCATIONS:
Overall Officials: Torng Pao-Ling, MD, PhD, Principal Investigator — Department of Obstetric and Gynecology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan